CLINICAL TRIAL: NCT01965561
Title: Performance of Junctional Tourniquets in Normal Human Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: United States Army Institute of Surgical Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, John F. Kragh, Jr, MD, Orthopedic Surgeon, Researcher, United States Army Institute of Surgical Research
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H-13-016
Record Dates: First submitted 2013-10-15; First posted 2013-10-18 (Estimated); Results first posted 2015-10-07 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CRoC (Experimental): Use of Combat Ready Clamp (CRoC)
  Interventions: Device: CRoC
- AAJT (Experimental): Use of Abdominal Aortic and Junctional Tourniquet
  Interventions: Device: AAJT
- JETT (Experimental): Junctional Emergency Treatment Tool
  Interventions: Device: JETT
- SJT (Experimental): SAM Junctional Tourniquet
  Interventions: Device: SJT

INTERVENTIONS:
Device: CRoC — Use of Combat Ready Clamp (CRoC)
  Arms: CRoC
Device: AAJT — Use of Abdominal Aortic and Junctional Tourniquet (AAJT)
  Arms: AAJT
Device: JETT — Use of Junctional Emergency Treatment Tool (JETT)
  Arms: JETT
Device: SJT — Use of SAM Junctional Tourniquet (SJT)
  Arms: SJT

SUMMARY:
Normal human adult volunteers wereused to investigate the performance of medical devices intended to stop junctional bleeding on the battlefield.

DETAILED DESCRIPTION:
Four FDA-cleared junctional tourniquets (Combat Ready Clamp (CRoC), Abdominal Aortic and Junctional Tourniquet (AAJT), Junctional Emergency Treatment Tool (JETT), and SAM Junctional Tourniquet (SJT)) wereassessed in a laboratory on healthy human volunteers. Lower extremity pulses were measured in 10 volunteers before and after junctional tourniquet application aimed at stopping the distal pulse assessed by Doppler auscultation. Tourniquets were applied in a randomized fashion, with 5 min rest periods between each application. Each tourniquet was applied to each subject, such that the subjects acted as their own controls.

ELIGIBILITY:
Inclusion Criteria:

* Adult human volunteers who are recruited, screened, and consent to participate
* Ages at least 18 years old to no more than 60 years old (<61) on the date of consent
* Male or female
* A worker for the US Military or US Government (active duty military, civilian employees, contractors)

Exclusion Criteria:

* Active-duty military subjects without their supervisor's permission to participate
* Detainees or prisoners
* Evidence of major disease of an artery (e.g., artery or vein surgery, atherosclerotic disease diagnosis, stroke, peripheral vascular disease or dysfunction such as Reynaud's phenomenon, migraine headaches, or cardiovascular disease [uncontrolled hypertension, heart attack, or arrhythmias]), active abdominal, inguinal, gluteal, or thigh disease, major deformity, or hernias
* Pregnancy
* Contracted employees to the US Military or US Government without contractual permission to participate in the research

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John F Kragh, MD, Principal Investigator — United States Army Institute of Surgical Research
Locations (1):
- United States Army Institute of Surgical Research, Forts Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Junctional Tourniquet Use: Junctional tourniquet use followed by rest, repeat. Rest = 5 minutes. SJT is belt with discs that inflate. JETT is belt with pads that screw down. AAT is a bladder within a belt. CRC is a vice.
Period: Overall Study
Arm/Group | Junctional Tourniquet Use
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Healthy human volunteers
Groups:
- Junctional Tourniquet Use: Junctional tourniquet use followed by rest, repeat
  Rest = 5 minutes. SJT is belt with discs that inflate. JETT is belt with pads that screw down. AAT is an bladder within a belt. CRC is a vice.
Arm/Group | Junctional Tourniquet Use
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] — Age of healthy human volunteers
  years | 51 [42 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Pain [Mean (Full Range); unit: units on a scale] — Pain level on Visual Analog Scale (0 mm = no pain, 100 mm = maximum pain)
  units on a scale | 0 [0 to 0]

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness at Stopping Distal Pulse
Description: Percentage of participants whose distal pulse ceased within 1 minute of junctional tourniquet application.
Time Frame: 1 min
Measure: Number; unit: percentage of participants
Groups:
- SJT Tourniquet: SAM Junctional Tourniquet (SJT)
Arm/Group | CRoC | AAJT | JETT | SJT Tourniquet
Number analyzed (Participants) | 10 | 10 | 10 | 10
percentage of participants | 97 | 27 | 83 | 93

2. Secondary Outcome: Pain During Tourniquet Application
Description: Pain during tourniquet application as measured on a visual analog scale (VAS). The pain scale was a 100-mm-long line on a piece of paper. The subject made a cross mark on the line, which went from the left limit (0 mm) at no pain to the right limit (100 mm) at very severe pain.
Time Frame: 1 minute
Measure: Mean (Standard Deviation); unit: mm on VAS
Arm/Group | CRoC | AAJT | JETT | SJT Tourniquet
Number analyzed (Participants) | 10 | 10 | 10 | 10
mm on VAS | 30 (23) | 76 (14) | 45 (40) | 43 (31)

ADVERSE EVENTS:
Groups:
- Junctional Tourniquet Use: Junctional tourniquet use followed by rest, repeat.
Arm/Group | Junctional Tourniquet Use
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes